CLINICAL TRIAL: NCT00147563
Title: A Double-Blind, Parallel Design Study to Compare the Effectiveness of Eplerenone Versus Atenolol in Reversing the Remodeling of Resistance Arteries in Subjects With Mild to Moderate Primary Hypertension
Brief Title: Compare Effectiveness of Eplerenone vs Atenolol in Reversing the Remodelling Resistance Arteries in Subjects With HT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPLA-0501-077; A6141016; NCT00260845 (obsolete NCT alias)
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2007-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Eplerenone

INTERVENTIONS:
Drug: Eplerenone

SUMMARY:
To investigate the impact of antihypertensive therapy with the selective mineralocorticoid receptor blocker, eplerenone, on small resistance artery remodeling, compared to the effect of equivalent blood pressure control achieved with a b-blocker, atenolol.

ELIGIBILITY:
Inclusion Criteria:

* Pt with essential hypertension who have never been treated or untreated within the previous 6 months

Exclusion Criteria:

* History of Malignant Hypertension
* Sitting diastolic blood pressure > 115mmHg or sitting Systolic blood pressure > 200mmHg

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34
Dates: Start 2003-10; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The change from baseline to week 52 in the media/lumen ratio and the maximum % relaxation response to acetylcholine of gluteal subcutaneous resistance vessels, measured from the gluteal biopsy.

SECONDARY OUTCOMES:
Will be done for both the Intent to Treat and per protocol populations, and use both the LOCF and OC methods

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Savoia C, Touyz RM, Amiri F, Schiffrin EL. Selective mineralocorticoid receptor blocker eplerenone reduces resistance artery stiffness in hypertensive patients. Hypertension. 2008 Feb;51(2):432-9. doi: 10.1161/HYPERTENSIONAHA.107.103267. Epub 2008 Jan 14. PMID 18195160
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=EPLA-0501-077&StudyName=Compare+effectiveness+of+Eplerenone+vs+Atenolol+in+reversing+the+remodelling+resistance+arteries+in+subjects+with+HT